CLINICAL TRIAL: NCT01573741
Title: Department of AnesthesiologyJinling Hospital, Nanjing University School of Medicine, Nanjing, China
Brief Title: Study of Ketamine as an Antidepressant in Major Depressive Disorder
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Jinyun (Other)
Responsible Party: Sponsor-Investigator, Shi Jinyun, Department of Anesthesiology, School of Medicine, Jinling Hospital, Nanjing, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: nju-030614
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder
Keywords: depressive ketamine antidepressant
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ketamine,four hours monitoring hydrochloride injection (Experimental): a single infusion of ketamine hydrochloride (0.5 mg/kg) infused over 40 minutes
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — a single infusion of ketamine hydrochloride (0.5 mg/kg) infused over 40 minutes

SUMMARY:
Primary Outcome Measures:

Evaluate the changes in neuroimaging and biochemistry measures with ketamine treatment.

Secondary Outcome Measures:

Evaluate the effects of ketamine on depression symptoms, manic symptoms, global change in psychiatric symptoms, and suicidal ideation.

ELIGIBILITY:
Inclusion Criteria:Male patients, ages 18 to 65 years with a diagnosis of MDD, currently depressed or in a current major depressive episode of BD without psychotic features will be recruited into this substudy.

Current or past history of lack of response to one adequate antidepressant trial, operationally defined using the Antidepressant Treatment History Form (ATHF); a failed adequate trial of ECT would count as an adequate antidepressant trial.

Exclusion Criteria:Subjects with a history of DSM-IV drug or alcohol dependency or abuse (except for caffeine or nicotine dependence) within the preceding 3 months. In addition, subjects who currently are using oher antidepressant drugs in the 2 weeks prior to screen and must have a negative alcohol and drug urine test (except for prescribed benzodiazepines) urine test at screening.

Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.

Presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications.

Clinically significant abnormal laboratory tests.

Subjects with clinical hypothyroidism or hyperthyroidism.

Subjects with one or more seizures without a clear and resolved etiology.

Presence of metallic (ferromagnetic) implants (e.g, heart pacemaker, aneurysm clip).

Subjects who, in the investigator's judgment, pose a current serious suicidal or homicidal risk, or who have a MADRS item 10 score

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
all cause remission | 7day
  Evaluate the effects of ketamine on depression symptoms, manic symptoms, global change in psychiatric symptoms, and suicidal ideation by MADRS,HDRS and SSI.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Yang, Dr, Study Chair — Department of Anesthesiology, Jinling Hospital, School of Medicine, Nanjing University
Locations (1):
- The PLA 102nd Hospital and mental health center of military, Changzhou, Jiangsu, China